CLINICAL TRIAL: NCT04378192
Title: Assessment of the Use of Laryngeal Mask Airway as Abridge for Intubation of Morbidly Obese Patients Undergoing Sleeve Gastrectomy
Brief Title: Laryngeal Mask Airway as a Bridge for Intubation of Obese Patients for Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LMA obesity
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Laryngeal Masks; Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face mask ventilation (Active Comparator): Use of face mask ventilation technique after induction of anaesthesia and administration pf muscle relaxant till the insertion of the endotracheal tube in a morbidly obese patient undergoing sleeve gastrectomy
  Interventions: Device: face mask
- Laryngeal mask ventilation (Active Comparator): Use of laryngeal mask airway LMA for ventilation after induction of anaesthesia and administration pf muscle relaxant till the insertion of the endotracheal tube in a morbidly obese patient undergoing sleeve gastrectomy
  Interventions: Device: Laryngeal mask airway

INTERVENTIONS:
Device: Laryngeal mask airway — Insertion of laryngeal mask airway before intubation of a morbidly obese patient
  Other Names: LMA
  Arms: Laryngeal mask ventilation
Device: face mask — use of face mask before intubation of a morbidly obese patient
  Arms: Face mask ventilation

SUMMARY:
Ventilation, as well as intubation of a morbidly obese patient, is challenging and require special preparations and skilful hands, in this study laryngeal mask airway insertion is used as a bridge for intubation to facilitate ventilation as give enough time to anaesthetics and muscle relaxants to work on.

DETAILED DESCRIPTION:
The ordinary pathway of intubating a morbidly obese patient for sleeve gastrectomy is bordered by the risk of difficult ventilation and intubation with the subsequent events of hypoxia and hypoventilation. When the patient is easy ventilated, it gives some sort of confidence and pleasure for the anaesthetist that the way of intubation will not be so hard.

One problem here is the difficulty of ventilating a morbidly obese patient, in this study the investigators used laryngeal mask airway as a bridge before inserting the endotracheal tube

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese patient BMI>40
* ASA I, II, III
* Elective sleeve gastrectomy

Exclusion Criteria:

* Oral cavity infection or pathological abnormalities
* Suspected or known abnormalities in supraglottic anatomy
* Patients planned for awake fiberoptic intubation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Time to intubation TTI | During the action of intubation after induction of anaesthesia
  The time starts with insertion of glidescop and ends at its withdrawal

SECONDARY OUTCOMES:
View of the glottis | During the action of intubation after induction of anaesthesia
  Based on the percentage of glottic opening (POGO) score as well as Cormack and Lehane's (C&L) classification
Number of attempts required for intubation, | During the action of intubation after induction of anaesthesia
  How many times the anaesthetist needs to try to succeed in insertion of the endotracheal tube
Anaesthetist's satisfaction score | During the action of intubation after induction of anaesthesia
  On a scale rang from 0 representing totally dissatisfied to 10 representing fully satisfied
Intubation difficulty score (IDS) | During the action of intubation after induction of anaesthesia
  Intubation difficulty score (IDS) is the sum of seven variables, each presents 1 point, score 0 represents easy intubation, score 1 to 5 represents moderate difficulty and score more than 5 was considered difficult intubation.
Need for external pressure during intubation | During the action of intubation after induction of anaesthesia
  to direct the larynx downward to facilitate endotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No